CLINICAL TRIAL: NCT06302309
Title: 'Managing the Mental State' to Tackle Anxiety-related Freezing of Gait in People With Parkinson's Disease: a Randomized Controlled Intervention Trial
Brief Title: Tackling Anxiety-related Freezing of Gait in People With Parkinson's Disease
Acronym: TACKLING-FOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL85217.091.23
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-03

CONDITIONS: Freezing of Gait
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Masking Description: Randomization will be performed in CastorEDC, a web-based data management system for academic studies (www.castoredc.com). Breaking of the randomization code is not applicable, since researchers and trainers cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive 4 sessions of the 'managing the mental state' intervention immediately after randomization.
  Interventions: Other: Psychological intervention
- Waitlist (Experimental): The control group will enter a waiting period of 4 weeks and receive the same 4-week intervention thereafter.
  Interventions: Other: Psychological intervention

INTERVENTIONS:
Other: Psychological intervention — The intervention consists of four sessions of a 'managing the mental state' intervention, of which the first and second session will take place in the home-setting of the patient; the two remaining sessions will take place remotely. The sessions include psychoeducation on what anxiety is and how stress and anxiety can influence FOG, identifying how people are allocating attention and engage in specific thought-processes (e.g. worrisome thoughts) during walking, and educating patients about 'managing the mental state' compensation strategies that involve ways to reduce anxiety or stress and will be specifically tailored to the individual patient.

SUMMARY:
The purpose of this study is to investigate whether personalized strategies that target anxiety and stress surrounding freezing of gait can alleviate freezing of gait in people with Parkinson's Disease.

DETAILED DESCRIPTION:
Rationale:

Freezing of Gait (FOG) is a common and disabling symptom in people with Parkinson's Disease (PD), characterized by paroxysmal episodes where there is an inability to step effectively, despite attempting to do so. Treatment consists of complementary pharmacological and non-pharmacological treatment options which unfortunately only partially alleviate FOG. Anxiety has been found to contribute to the occurrence and exacerbation of FOG, which often manifests itself in situations where people with FOG anticipate not being in control of their movements. People with FOG are often aware of the feelings and situations that elicit FOG episodes, but they rarely actively employ strategies targeting their mental state to improve FOG. With the exception of general interventions including mindfulness, yoga and meditation, tailored strategies to ameliorate anxiety-related FOG have never been evaluated in a systematic manner.

Objective:

In this project we aim to evaluate whether a non-pharmacological and tailored intervention targeting anxiety- and stress-related FOG in people with PD is effective to reduce the impact of anxiety and stress on FOG. Specifically, we aim to study: (1) the effect of four sessions of a 'managing the mental state' intervention in people with disabling and anxiety-related FOG; and (2) the key determinants of the effectiveness of the intervention to reduce the impact of anxiety and stress on FOG.

Study design:

This study is a randomized controlled trial (RCT). The intervention group will receive the intervention immediately after randomization while a (waitlist) control group receives the same intervention thereafter.

Study population:

Forty people with PD that experience daily FOG (as objectified with the new-freezing of gait questionnaire) will be included, that is related to anxiety (positive answer to the question: Does FOG occur or get worse when you are anxious or stressed?).

Intervention:

The intervention consists of four sessions of a 'managing the mental state' intervention, of which the first and second session will take place in the home-setting of the patient; the two remaining sessions will take place remotely. The sessions include psychoeducation on what anxiety is and how stress and anxiety can influence FOG, identifying how people are allocating attention and engage in specific thought-processes (e.g. worrisome thoughts) during walking, and educating patients about 'managing the mental state' compensation strategies that involve ways to reduce anxiety or stress and will be specifically tailored to the individual patient.

Main study parameters/endpoints:

The primary outcome involves the percentage of time frozen during a home-based gait trajectory with self-selected FOG 'hotspots'. Secondary outcomes involve the subjective impact of anxiety and stress on FOG, as measured with a Visual Analogue Scale and the perceived levels of anxiety.

ELIGIBILITY:
Inclusion Criteria:

Men/women of age > 18 years with idiopathic Parkinson's disease, as diagnosed by the UK Brain Bank Criteria;

* Presence of daily FOG (as objectified with the new-freezing of gait questionnaire), that is related to anxiety (positive answer to the question: Does FOG occur -or get worse when you are anxious or stressed?);
* Using a stable dose of PD medication and stability of DBS settings (if applicable) during the trial. Adjustments of PD medication and DBS settings during the trial are allowed if deemed clinically necessary.
* Written informed consent.

Exclusion Criteria:

* Any comorbidity (i.e. neurological, orthopedic) that significantly impacts gait.

  * Severe cognitive impairment hampering the ability to comply to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
% time frozen during a personalized gait trajectory | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The primary outcome measure involves the percentage of time frozen during a personalized walking trajectory that includes self-selected FOG 'hotspots' in the home setting. This gait trajectory will be exactly the same during the baseline and consecutive measurements, and will be performed at comfortable gait speed. The gait trajectory will be video-taped by the assessor and performed three times during each visit.

SECONDARY OUTCOMES:
subjective impact of anxiety and stress on FOG, as measured with a Visual Analogue Scale | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  subjective impact of anxiety and stress on FOG, as measured with a Visual Analogue Scale
Heart Rate Variability | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  Heart rate variability (HRV) will be measured to determine whether the gait measures induce physiological stress and to examine if the intervention leads to a reduction in physiological stress. For this purpose, we will collect 3-lead electrocardiogram signals for heart rate monitoring prior to and during the gait measures
The Parkinson Anxiety Scale (PAS) | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Parkinson Anxiety Scale (PAS) [9] is a questionnaire that has been specifically developed for measuring anxiety in people with PD.
Gait-Specific Attention Profile | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Gait-specific attentional profile (G-SAP) provides measurements of multiple psychological factors that influence gait performance. The G-SAP will be administered in order to determine whether psychological factors that are implicated in gait performance (e.g., conscious processing of movement, fall-related ruminations) are changed in response to the intervention
he Updated Perceived Control over Falling Scale (UP-COF) | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Updated Perceived Control over Falling Scale (UP-COF) is a 4-item scale that will be administered to assess whether the intervention improves participants' perceived control over the risk of falling.
New Freezing of Gait Questionnaire | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The New-Freezing of Gait Questionnaire (N-FOGQ) assesses the subjective severity of Freezing of Gait.
The Parkinson's Disease Questionnaire | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Parkinson's Disease Questionnaire (PDQ-39) will be administered to measure quality of life.
The Rosenberg self-esteem score | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Rosenberg self-esteem score will be administered in order to assess self-esteem.
Perceived Stress Scale | Baseline, week after the intervention has ended (5 weeks from baseline) and 10 week follow-up (15 weeks from baseline)
  The Perceived Stress Scale will be administered in order to determine whether the intervention leads to a decrease in perceived levels of stress.

OTHER OUTCOMES:
Montreal Cognitive Assessment | Baseline
  The Montreal cognitive assessment will be measured at baseline to determine cognitive status
Unified Parkinson's Disease Rating Scale Part III | Baseline
  Part III of the UPDRS is a physical examination that examines the severity of Parkinson's Disease motor symptoms. The UPDRS will be administered at baseline to measure Parkinson's Disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Jorik Nonnekes, PhD, Principal Investigator — Radboud University Medical Center (Radboudumc)
Locations (1):
- Department of Rehabilitation Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No